CLINICAL TRIAL: NCT00578994
Title: A Prospective, Non-randomized, Multicenter Study of the Oxford® Meniscal Unicompartmental Knee System
Brief Title: A Clinical Investigation of the Oxford® Meniscal Unicompartmental Knee System
Status: Completed | Type: Observational
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: ORTHO.CR.K016; P010014 (Other: FDA PMA)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis; Avascular Necrosis
Keywords: Unicompartmental Knee; Partial Knee; Knee arthroplasty
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Oxford® Meniscal Unicompartmental Knee: Patients with PKA using the Oxford® Meniscal Unicompartmental Knee System
  Interventions: Device: Oxford® Meniscal Unicompartmental Knee System

INTERVENTIONS:
Device: Oxford® Meniscal Unicompartmental Knee System — Oxford® Meniscal Unicompartmental Knee System is a medial, unicompartmental knee prosthesis containing three components: a femoral component, a tibial component, and a tibial meniscal bearing.

SUMMARY:
The purpose of this study is to collect information on complications and survivorship of patients implanted with the Oxford™ Meniscal Unicompartmental Knee System at multiple sites in the United States.

DETAILED DESCRIPTION:
Study Objective

To provide a prospective 2-year post-operative evaluation of complications and 9-year long-term survivorship analysis of patients implanted with the Oxford™ Meniscal Unicompartmental Knee System at multiple sites in the United States.

Study Design

The study is designed as a prospective, multi-center, non-randomized post approval study. There are two phases to this study:

1. A complications study where patients will be followed for at least 2 years to record all complications that may occur, and
2. A survival study that will record at yearly intervals out to 9 years whether or not the device is still in place or if it has been removed for any reason.

Phase 1 requires clinical follow-up (0-2 year) and patients will be evaluated at pre-defined intervals up to 2 years post-operative. Information gathered in phase 1 includes all adverse events and survival data.

Phase 2 (3-9 year) only gathers survival data through patient directed mailing and/or phone call.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of the following diagnoses in the medial compartment of the knee: Osteoarthritis, Avascular Necrosis

Exclusion Criteria:

* Patients with Rheumatoid arthritis or other forms of inflammatory joint disease
* Patients with infection, sepsis, and osteomyelitis
* Patients with Osteoporosis, Paget's Disease, Charcot's disease, Osteomalacia, and Severe Osteoporosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A Multi-center study conducted in the United States of patients who meet the FDA approved indications for use. The Oxford Meniscal Unicompartmental Knee System is intended for use in individuals with osteoarthritis or avascular necrosis limited to the medial compartment of the knee and is intended to be implanted with bone cement.
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2006-03; Primary Completion 2019-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Survivorship | Annually for 9 years post-op
  Assessment of frequency of Revisions

SECONDARY OUTCOMES:
Complications | 2 Years
  Patients will be followed for at least 2 years to record all complications that may occur

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, Study Director — kacy.arnold@zimmerbiomet.com
Locations (6):
- United States (6):
  - Barrington Orthopedic Specialissts, Schaumburg, Illinois
  - Joint Implant Surgeons, New Albany, Ohio
  - Mid-South Orthopedic Associates, Cordova, Tennessee
  - Texas Orthopedic Specialist, Bedford, Texas
  - Texas Center for Joint Replacement, Plano, Texas
  - Advanced Orthopaedic Centers, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided